CLINICAL TRIAL: NCT05261321
Title: Cannabis and Polysubstance Use: Response Inhibition and Stress Exposure
Acronym: CAPU RISE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christian Schutz, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CAPU RISE 1.0
Record Dates: First submitted 2022-01-25; First posted 2022-03-02 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: cannabis; cannabinoids; stress; neuroimaging; fMRI
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded masking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cannabis oil with a high ratio of THC to CBD (Active Comparator): Participants will be given a single dose of oral cannabis oil containing 5mg THC and 0.17mg CBD.
  Interventions: Drug: Cannabis oil with a high ratio of THC to CBD
- Cannabis oil with a high ratio of CBD to THC (Active Comparator): Participants will be given a single dose of oral cannabis oil containing 5mg THC and 25mg CBD.
  Interventions: Drug: Cannabis oil with a high ratio of CBD to THC
- Placebo (Placebo Comparator): Participants will be given a single dose of 1 mL placebo (carrier oil with botanical terpenes) via oral route of administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabis oil with a high ratio of THC to CBD — In the first active condition, cannabis oil with a high THC to CBD ratio will be administered to participants.
  Arms: Cannabis oil with a high ratio of THC to CBD
Drug: Cannabis oil with a high ratio of CBD to THC — In the second active condition, cannabis oil with a high CBD to THC ratio will be administered to participants.
  Arms: Cannabis oil with a high ratio of CBD to THC
Drug: Placebo — In the control condition, the placebo will be administered to participants.
  Arms: Placebo

SUMMARY:
The purpose of this Phase I non-therapeutic trial is to examine the neurological effects of cannabis on stress reactivity and inhibition in healthy cannabis users. We expect differences between high ratio CBD:THC cannabis oil, low ratio CBD:THC cannabis oil, and/or placebo on outcome measures.

DETAILED DESCRIPTION:
Purpose: To examine the neurological effects of cannabis on stress reactivity and inhibition in healthy adults using recreational cannabis. This is a phase I/pilot healthy subjects trial.

Primary Hypotheses:

1. The intervention will be feasible to implement
2. Cannabis oil will attenuate stress, measured via biological and self-report data, including salivary molecules, functional Magnetic Resonance Imaging, and standardized psychosocial assessments.

Justification: Current cannabis research focuses on medical uses for cannabis, clinical populations and/or non-commercially available products. There remains limited experimental research on the effects of commercial products in non-clinical regular users of cannabis. Further, most drug use research excludes polysubstance users. Given the high number of people using cannabis to cope with stress, biological evidence is needed to determine the validity of this claim. Stress is known to negatively impact daily functioning and has been linked to poorer mental and physical health outcomes. The effects of cannabinoids on cognitive functioning also have implications for daily functioning.

Objectives: Determine a causal link between commercially available cannabinoid products and mechanisms involved with stress response in polysubstance users, specifically weekly cannabis users with heavy drinking (males: minimum 5 drinks, females: minimum 4 drinks on at least one occasional per month for the past 12 months). Examine the short-term effects of cannabinoids on sleep quality in this population.

Study Design: The study is a Phase I non-therapeutic pilot trial and will utilize a double-blind, placebo-controlled, within-subjects design. The acute effects of the investigational products (IPs) will be examined. Each participant will undergo an initial phone screen and 5 sessions, with sessions 2-4 involving drug administration. There will be three investigational product arms for the drug administration sessions: cannabis oil with a high ratio of THC to CBD, cannabis oil with a high ratio of CBD to THC, and placebo. Each participant will be exposed to all three arms, one per drug administration session. The order of arm will be randomized. Each drug administration session will be a minimum of10 days apart to ensure a sufficient washout period.

ELIGIBILITY:
Inclusion criteria:

1. Are 19-35 years old at the start of the study
2. Have used oral cannabis for non-medical purposes twice the past month (30 days)
3. Have previously used a minimum of 20mg of CBD
4. Have previously used a minimum of 5mg THC
5. Are using an effective and/or highly effective method of contraception and will continue to do so for the duration of participation in the study. Health Canada's definition of effective methods of contraception include barrier methods of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge). Health Canada's definition of highly effective methods of contraception includes hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy and tubal ligation.
6. Females: are not undergoing alternative fertility methods, such as IVF, or otherwise trying to start a family for the duration of participation
7. Males: will not be donating sperm at some point during the duration of participation
8. Are able to provide informed consent
9. Are able to complete assessments in English
10. Are able to attend sessions according to the study schedule
11. Will provide proof of 2 doses of an approved COVID-19 vaccination

Exclusion criteria:

1. Are left-handed or ambidextrous
2. Females: are pregnant, nursing, or not on safe pregnancy protection
3. Are trying to conceive
4. Have a known or suspected allergy to cannabinoids and/or palm/coconut oil
5. Are hypersensitive to CBD and/or THC and/or have ever had an adverse reaction (an unwanted and unexpected reaction), to less than 40mg of CBD and/or 10mg THC
6. Have had an adverse reaction (unwanted, unexpected reaction or symptoms) to cannabis within last 6 months
7. Have a major physical problem/health concern, including:

   1. Liver-cirrhosis or other liver disease
   2. Diabetes
   3. Chronic illness that may increase risk for adverse reactions to cannabis
   4. Chronic pain
   5. Genetic glucuronidation disorders (e.g., Gilbert's disease)
   6. Cardiovascular disease, including ischemic heart disease with unstable angina or recent acute coronary syndrome in the last 3 months, uncontrolled arrhythmias, poorly controlled hypertension or high blood pressure (e.g., 130/80), or severe heart failure
   7. Delirium: active delirium or recent delirium < 7 days, or at significant risk of delirium due to multiple comorbidities (e.g., very elderly, cognitive impairment, cerebrovascular disease) and contributing drugs (e.g., alcohol, stimulants, high doses of benzodiazepines, opioid, sedatives, psychoactive medications)
8. Are taking any of the following medications:

   1. Any medication that impacts the central nervous system, brain, and/or metabolic system
   2. Psychotropic medications, sedatives, and central nervous system depressants, including sleeping pills, tranquilizers, some pain medications, some allergy and cold medications, and anti-seizure medications
   3. Medications otherwise affecting the central nervous system, including amphetamines and other sympathomimetics
   4. Allergy medications (antihistamines; within 24 hours)
   5. Heart medications
   6. Blood pressure medication
   7. Steroid medications
   8. Opioids or other pain medications
   9. Anticholinergics: drugs that block acetylcholine, a chemical signal that plays a role in memory and learning.
   10. Drugs metabolized by cytochrome P450 enzymes, including amitriptyline, fentanyl, sufentanil, and alfentanil
   11. Highly protein-bound drugs, including warfarin, cyclosporine, and amphtericin
   12. Drugs metabolized by UGT enzymes, including propofol, antivirals
   13. Antiretroviral drugs
   14. Stomach acid inhibitors
   15. Antibiotics and antifungal medications
   16. Heart medications
   17. Other medications/substances interfering with CYP2C19 receptors

   i. Inhibitors: Fluvoxamine, isoniazid (INH), ritonavir ii. Inducers: Carbamazepine, phenytoin, rifampin iii. Substrates: Omeprazole (Prilosec), phenobarbital, phenytoin r. Other medications/substances interfering with CYP3A4 receptors: i. Inhibitors: Clarithromycin (Biaxin), diltiazem (Cardizem), erythromycin, grapefruit juice, itraconazole (Sporanox), ketoconazole (Nizoral), nefazodone (Serzone), ritonavir, telithromycin (Ketek), verapamil (Calan) ii. Inducers: Carbamazepine, Hypericum perforatum (St. John's wort), phenobarbital, phenytoin, rifampin iii. Substrates: Alprazolam (Xanax), amlodipine (Norvasc), atorvastatin (Lipitor), cyclosporine (Sandimmune), diazepam (Valium), estradiol (Estrace), simvastatin (Zocor), sildenafil (Viagra), verapamil, zolpidem (Ambien)
9. Other MRI contraindications (conditions that make MRI procedure inadvisable):

   a. Have implanted metal clips or wires, including: i. Implanted electronic device (e.g., pacemaker, defibrillator implanted medication infusion pump, electrical stimulator, and/or ear or eye implant) including retained wires that has been removed (e.g., pacemaker wires not attached to a pacemaker) ii. Stainless steel intrauterine device (IUD) iii. Metal in eye or orbit, or metal slivers iv. Ferromagnetic aneurysm clip v. Coil, catheter, or filter in any blood vessel vi. Orthopedic hardware (artificial joint, plate, screw, rod) vii. Shrapnel, bullets, or other metal fragments (i.e., metal in eye or orbit) viii. Artificial heart valve ix. Ear or eye implant x. Brain aneurysm clip xi. Implanted electronic device (i.e., drug infusion pump, electrical stimulator) xii. Coil, catheter, or filter in any blood vessel xiii. Surgery, medical procedure or tattoos (including tattooed eyeliner) in the last six weeks xiv. Other metallic prostheses b. Have a personal or family history of seizures c. Have any significant neurological disorder including, but not limited to: i. Any condition likely to be associated with increased intracranial pressure ii. Space-occupying brain lesion iii. Seizure iv. Cerebral aneurysm v. Parkinson's disease vi. Huntington's chorea vii. Multiple sclerosis viii. Significant head trauma with loss of consciousness for greater than or equal to 5 minutes d. Claustrophobia (i.e., feel uncomfortable in small spaces) or fear of loud, repetitive sounds, or inability to lay still. Participants will have to lie still in the confined space of the MRI scanner.
10. Work nightshifts
11. Have any diagnosed sleep disorders
12. Have dyscalculia
13. Have a neurodevelopmental disorder or cognitive impairments, including:

    1. Autism Spectrum Disorder
    2. Attention Deficit/Hyperactivity Disorder (ADHD)
14. Have schizophrenia spectrum disorder and/or history of psychosis
15. Meet criteria for potential mental health disorder in the Mini International Neuropsychiatric Interview (M.I.N.I.) Screen Version 7.0.2, except for alcohol and cannabis use disorders
16. Any diagnosed current mental health disorder and/or diagnosis of a mental health disorder within the past year
17. Have a non-correctable clinically significant sensory impairment (e.g., cannot hear well enough to cooperate with interview)

19) Are unable to attend sessions according to the study schedule 20) Have used opiates more than twice in the past 30 days

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in stress response across conditions | 5 weeks
  Indicated by differences in blood-oxygenation-level-imaging (BOLD) response via functional magnetic resonance imaging (fMRI), salivary stress molecule levels (eg cortisol, IgA), heart rate, and self-reports. Participants will fill out a daily diary each morning starting the day after session 1 until the day of session 5 with their self-reports.
Change in incidence of adverse events of cannabinoids across conditions | 5 weeks
  Assessed through self-reports from study participants (semi-structured interviews) and clinically significant adverse changes in vital signs (heart rate, blood pressure).
Procedure feasibility | Through study completion; average of 1 year
  Measured via means and rates of study recruitment
Protocol feasibility | Through study completion; average of 1 year
  Measured via means and rates of study recruitment

SECONDARY OUTCOMES:
Change in performance on behavioral impulsivity tasks across conditions | 5 weeks
  Measured by Delay and Probability Discounting Procedure, Experiential Discounting Task, and the Hybrid Response Inhibition Task
Change in sleep quality across conditions | 5 weeks
  Measured via wrist-worn actigraphy using the Fatigue Science Readiband and self-report based on the Pittsburgh Sleep Inventory
Change in subjective response to cannabis | 5 weeks
  Measured via Drug Effects Questionnaire, assessing aspects of subjective response on a scale from "Not at All" to "Extremely", "Dislike Very Much" to "Like Very Much", and other variations.
Change in state anxiety across conditions | 5 weeks
  Measured by State Anxiety sub-scale of the State Trait Anxiety sub-scale, rating experience from "Not at All" to "Very Much"
Change in psychological distress across conditions | 5 weeks
  Measured by the standardized Short Form of the Profile of Mood States, assessing experience of various feelings from "Not at All" to "Extremely"

CONTACTS AND LOCATIONS:
Overall Officials: Christian G Schütz, MD PhD, Principal Investigator — University of British Columbia; British Columbia Mental Health and Substance Use Services; Karina A Thiessen, BA BEd, Study Director — University of British Columbia
Locations (1):
- B.R.A.I.N. Lab, Institute of Mental Health, Faculty of Medicine, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No